CLINICAL TRIAL: NCT01315769
Title: COMPARATIVE STUDY OF PELVIC FLOOR MUSCLE EVALUATION IN NULIPAROUS AND PRIMIPAROUS WOMEN. A Prospective Study
Brief Title: Pelvic Floor Muscle Function in Nulliparous and Primiparous.
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Prof. Trajano Sardenberg, Ethical Research Committee
Other Study IDs: upeclin/HC/FMB-Unesp-51
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Investigation or Care in A Nonpregnant Woman; Mother (Person)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non pregnant nulliparous: Group 1
- primiparous women: Group 2

SUMMARY:
This study aimed to compare the pelvic floor muscle (PFM) strength in nulliparous and primiparous women. Subjective evaluation of PFM strength was performed vaginal digital palpation (TDP). The objective evaluation of PFM strength was assessed using a portable perineometer. All parameters were performed at one moment in G1, and in G2, during the 20th and 36th weeks of pregnancy, and 45 days after the delivery. Pregnancy and vaginal delivery may cause weakness of PFM.

DETAILED DESCRIPTION:
Objective: This study aimed to compare the pelvic floor muscle (PFM) strength in nulliparous and primiparous women. Populations: The sample size was established considering a significance level of 5%, the test power of 80%, and the estimated error of 10%. According to these results and considering the range between percentages of answers as the casual error, each group was established with approximately 50 participants. Methods: 100 women were prospectively distributed into: Group G1 (n = 50) comprising by healthy nulliparous women; Group G2 (n = 50) with primiparous ones. Subjective evaluation of PFM strength was performed using transvaginal digital palpation (TDP). The objective evaluation of PFM strength was assessed using a portable perineometer. All parameters were performed at one moment in G1, and in G2, during the 20th and 36th weeks of pregnancy, and 45 days after the delivery. Results: In G2, 14 women were excluded due to the lost follow-up. The median of age was 23 years in G1 and 22, in G2, there was no statistical difference between the groups. In G1, BMI was in average 21.7 Kg/m2, and 25,0 Kg/m2 in G2, there was statistical difference between the groups (p= 0.0004). In G2, TDP evaluation showed a significant impairment of PFM strength at 36th week of pregnancy (p=0,0006) and 45 days after the vaginal delivery (p=0.0001) compared to nulliparous. Objective evaluations of PFM strength showed a significant decrease 45 days after vaginal delivery compared to nulliparas. Conclusion: Pregnancy and vaginal delivery may cause weakness of PFM.

ELIGIBILITY:
Inclusion Criteria:

- Nulliparous and primiparous

Exclusion Criteria:

* in G1 (nulliparous) were UI, neurological diseases, previous pelvic surgeries, diabetes, smoking and cognitive difficulties. In G2 (primiparas), the same criteria were used including women with gestational complications such as diabetes, hypertension, vaginal and urinary infection.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The sample size was established considering a significance level of 5%, the test power of 80%, and the estimated error of 10%. According to these results and considering the range between percentages of answers as the casual error, each group was established with approximately 50 participants.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-03; Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joao L Amaro, PhD MD, Principal Investigator — Urology Department
Locations (1):
- Medical School of Botucatu, Botucatu, São Paulo, Brazil